CLINICAL TRIAL: NCT07354464
Title: Efficacy of Sphenopalatine Block Compared to Blood Patch in the Management of Post-dural Puncture Headaches
Acronym: BRECHE
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RBHP 2025 GUYOT (BRECHE); 2025-522168-34-00 (EU CTIS Number)
Record Dates: First submitted 2026-01-07; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-11

CONDITIONS: PDPH; Post Dural Puncture Headache
Keywords: Post Dural Puncture Headache; Blood patch; Sphenopalatin ganglion block
MeSH Terms: conditions — Post-Dural Puncture Headache | interventions — Sphenopalatine Ganglion Block; Blood Patch, Epidural

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blood patch (Active Comparator): Clinicians perform an epidural blood patch following current clinical guidelines.
  Interventions: Drug: Blood patch
- Sphenopalatin ganglion block (Experimental): Clinicians perform a sphenopalatin ganglion block following current clinical guidelines.
  Interventions: Drug: Sphenopalatine Ganglion Block

INTERVENTIONS:
Drug: Sphenopalatine Ganglion Block — The sphenopalatine ganglion block is performed in the post-anesthesia care unit (PACU). The patient is continuously monitored, including measurement of oxygen saturation, heart rate, and arterial blood pressure. The patient is placed in the supine position with the head extended. The anesthesiologist inserts a cotton-tipped applicator (sterile microbiology swab) soaked with 2.5% lidocaine cream into each nasal cavity until bony contact is reached. Subsequently, 1 mL of 5% injectable lidocaine is administered into each nasal cavity. The cotton-tipped applicators are left in place for 10 minutes and then removed. If headache persists upon patient mobilization to the upright position, the sphenopalatine ganglion block may be repeated a second time.
  Arms: Sphenopalatin ganglion block
Drug: Blood patch — The epidural blood patch is performed in the post-anesthesia care unit (PACU). The patient is continuously monitored, with measurement of oxygen saturation, heart rate, and arterial blood pressure. The patient is seated at the edge of the bed, with the anesthesiologist positioned behind the patient. The procedure is carried out in strict adherence to aseptic techniques. The puncture is ideally performed at the L3-L4 or L4-L5 interspace, preferably at or below the level of the initial puncture. Local anesthesia is achieved using 1% injectable lidocaine at the puncture site. The epidural space is identified using the loss-of-resistance technique with saline. Once the epidural space has been identified, peripheral venous blood is collected and slowly injected into the epidural space until the patient reports a sensation of pressure or lumbar pain, with a maximum volume of 30 mL. The patient is then placed in the strict supine position and monitored for at least 30 minutes in the PACU.
  Arms: Blood patch

SUMMARY:
Post-dural puncture headache (PDPH) is an iatrogenic complication following a dural puncture, which may occur after lumbar puncture, spinal or epidural anesthesia. These headaches are defined as positional headaches, which worsen in the upright position and improve in the supine position, occurring within 5 days after a dural puncture.

PDPH is disabling, particularly in the postpartum period and is often associated with symptoms such as nausea, vomiting, neck stiffness, photophobia, and hearing loss. While serious immediate complications (e.g., subdural hematoma, cerebral venous thrombosis) are rare, long-term consequences - including chronic headaches, neck or low back pain and depression, have been described.

A conservative treatment is usually started during the first 24 hours, but it often proves insufficient, leading to the use of an additional epidural blood patch therapy. While considered as the gold standard, this procedure is invasive and presents limitations. The effectiveness of the epidural blood patch is variable (33-91 %), and the need for a second blood patch is not uncommon. The risks associated with the procedure include second dural puncture, low back pain, vasovagal syncope and paresthesia. Serious complications could occur with reported cases of aseptic meningitis or acute subdural hematoma.

An emerging alternative is the sphenopalatine ganglion block that is a less invasive procedure showing promising results. Several recent trials suggested the safety, feasibilty and efficacy of this intervention with excellent tolerance. Then, we aim to compare the efficacy and safety of these procedures in a randomized controlled trial.

DETAILED DESCRIPTION:
This is a single-center interventional study classified as a clinical drug trial (European Regulation n°536-2014).

Patients suffering from post-dural puncture headache resistant to medical treatment for 24 hours are refered by the treating physician to the referent anesthesia team for consultation.

Patient screening for the study is realised and study information is delivered by the anesthesia team. After the verification of inclusion and non-inclusion criteria, inform consent is searched. The patient is managed either with an epidural blood patch or a sphenopalatine ganglion block, depending on the group of randomisation. During at least 30 minutes post-intervention, patients are monitored in the post-anesthesia care unit.

Headache intensity is assessed using the numerical rating scale just before the intervention and at 30 minutes, 1 hour, 2 hours, 6 hours, 24 hours, 48 hours and 7 days post-intervention. All secondary outcomes are evaluated during the 7 days after the intervention. This assessment is carried out by a clinical research associate blinded to the treatment allocation.

The patient will be hospitalized for at least 6 hours and if the treatment is ineffective after 24 hours, a rescue therapy with an epidural blood patch will be mandated, regardless of the patient's randomization group. If the patient is discharged within 7 days follow up the intervention, the numerical rating scale and secondary outcomes assessments will be conducted by telephone.

ELIGIBILITY:
Inclusion Criteria:

* Patients with post-dural puncture headache meeting the criteria of the International Classification of Headache Disorders (ICHD-3) and persisting after 24 hours of conservative treatment,
* Patients aged over 18 years,
* Patients affiliated to a social security health insurance system,
* Patients who have provided written informed consent.

Exclusion Criteria:

* Patients under legal protection (guardianship or curatorship), deprived of liberty (prisoners), or under judicial safeguard,
* Pregnant patients,
* Patients with hypersensitivity to lidocaine, prilocaine, local anesthetics of the amide type, or to any of the excipients listed in the composition of the drugs used in the protocol,
* Patients with acute porphyria, atrioventricular conduction disorders requiring permanent cardiac pacing not yet implemented, or epilepsy not controlled by treatment,
* Patients receiving antiarrhythmic therapy associated with torsades de pointes (amiodarone, disopyramide, quinidine derivatives, sotalol, etc.),
* Patients with atypical post-dural puncture headache suggestive of a post-dural puncture complication (altered consciousness, focal neurological deficit, seizures, visual disturbances, etc.),
* Patients with chronic headaches requiring preventive treatment,
* Patients with a history of spinal surgery precluding the performance of an epidural blood patch,
* Patients with contraindications to epidural blood patch (local or systemic infection, platelet count < 80 G/L, coagulation disorders, progressive neurological disease),
* Patients with contraindications to sphenopalatine ganglion block (nasal polyposis, rhinopharyngitis, deviated nasal septum).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
The main objective of our study is to evaluate the efficacy of the sphenopalatine ganglion block in the management of post-dural puncture headache compared to the epidural blood patch. | From the beginning of the intervention to the end of following at 7 days
  The primary outcome measure is the evolution of headache intensity in standing position, evaluated using a numerical rating scale [ranging from 0 (no pain) to 10 (the worst pain ever)] at the beginning of the intervention, at 30 minutes, 1 hour, 2 hours, 6 hours, 24 hours, 48 hours and 7 days after the performance of a sphenopalatine ganglion block or an epidural blood patch.

SECONDARY OUTCOMES:
The proportion of patients considered to be in pain | At 30 minutes, 1 hour, 2 hours, 6 hours, 24 hours, 48 hours, and 7 days
  Proportion of patients experiencing pain according to thresholds commonly reported in the literature and evaluated using a numerical rating scale [ranging from 0 (no pain) to 10 (the worst pain ever)]
Analgesic consumption | After the initial procedure to the end of following at 7 days
  Analgesic consumption (paracetamol, nefopam, NSAIDs, opioids) in milligrams after the procedure
The need for rescue therapy | After the initial procedure to the end of following at 7 days
  Need for rescue treatment with an epidural blood patch after the initial procedure
Length of hospital stay | From enrollment to the end of following at 7 days
Headache intensity at different time points | At 30 minutes, 1 hour, 2 hours, 6 hours, 24 hours, 48 hours, and 7 days post-intervention.
  Headache intensity is evaluated using a numerical rating scale [ranging from 0 (no pain) to 10 (the worst pain ever)]
Occurrence of adverse events | During the procedure
Occurrence of serious adverse events | From enrollment to the end of following at 7 days
Patient satisfaction | At day 7 post-intervention.
  Patient satisfaction assessed 7 days after treatment using a 5-item Likert scale.
  The Likert scale is a 5-point forced-choice scale (strongly agree, agree, neither agree nor disagree, disagree, strongly disagree). It is a widely used ordinal psychometric tool that assesses the degree of agreement or disagreement of respondents with a series of items. In this study, the following items were used:
  * The procedure (epidural blood patch or sphenopalatine ganglion block) was an unpleasant/painful experience.
  * The procedure (epidural blood patch or sphenopalatine ganglion block) effectively relieved my headache.
  * The procedure (epidural blood patch or sphenopalatine ganglion block) provided rapid relief of my headache.
  * At present, I no longer experience any symptoms of post-dural puncture headache.

CONTACTS AND LOCATIONS:
Overall Officials: Adrien Guyot, Principal Investigator — CHU de Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cohen S, Levin D, Mellender S, Zhao R, Patel P, Grubb W, Kiss G. Topical Sphenopalatine Ganglion Block Compared With Epidural Blood Patch for Postdural Puncture Headache Management in Postpartum Patients: A Retrospective Review. Reg Anesth Pain Med. 2018 Nov;43(8):880-884. doi: 10.1097/AAP.0000000000000840. PMID 30063655
- [Result] Gayathri GA, Karthik K, Saravanan R, Meshach MD, Pushparani A. A randomized control study to assess the efficacy of the sphenopalatine ganglion block in patients with post dural puncture headache. Saudi J Anaesth. 2022 Oct-Dec;16(4):401-405. doi: 10.4103/sja.sja_780_21. Epub 2022 Sep 3. PMID 36337388
- [Result] Dwivedi P, Singh P, Patel TK, Bajpai V, Kabi A, Singh Y, Sharma S, Kishore S. Trans-nasal sphenopalatine ganglion block for post-dural puncture headache management: a meta-analysis of randomized trials. Braz J Anesthesiol. 2023 Nov-Dec;73(6):782-793. doi: 10.1016/j.bjane.2023.06.002. Epub 2023 Jul 6. PMID 37422191
- [Result] Jespersen MS, Jaeger P, AEgidius KL, Fabritius ML, Duch P, Rye I, Afshari A, Meyhoff CS. Sphenopalatine ganglion block for the treatment of postdural puncture headache: a randomised, blinded, clinical trial. Br J Anaesth. 2020 Jun;124(6):739-747. doi: 10.1016/j.bja.2020.02.025. Epub 2020 Apr 15. PMID 32303377
- [Result] Kassim Z, Kamar RM, Zakariah MF, Chui Geok IS. Transnasal sphenopalatine ganglion block for postdural puncture headache in obstetric patients: A Malaysian experience report. J Taibah Univ Med Sci. 2022 Feb 25;17(5):805-809. doi: 10.1016/j.jtumed.2022.02.008. eCollection 2022 Oct. PMID 36050945
- [Result] Puthenveettil N, Rajan S, Mohan A, Paul J, Kumar L. Sphenopalatine ganglion block for treatment of post-dural puncture headache in obstetric patients: An observational study. Indian J Anaesth. 2018 Dec;62(12):972-977. doi: 10.4103/ija.IJA_443_18. PMID 30636799
- [Result] Cohen S, Trnovski S, Zada Y. A new interest in an old remedy for headache and backache for our obstetric patients: a sphenopalatine ganglion block. Anaesthesia. 2001 Jun;56(6):606-7. No abstract available. PMID 11412202
- [Result] Nair AS, Rayani BK. Sphenopalatine ganglion block for relieving postdural puncture headache: technique and mechanism of action of block with a narrative review of efficacy. Korean J Pain. 2017 Apr;30(2):93-97. doi: 10.3344/kjp.2017.30.2.93. Epub 2017 Mar 31. PMID 28416992
- [Result] Williams EJ, Beaulieu P, Fawcett WJ, Jenkins JG. Efficacy of epidural blood patch in the obstetric population. Int J Obstet Anesth. 1999 Apr;8(2):105-9. doi: 10.1016/s0959-289x(99)80007-7. PMID 15321154
- [Result] Booth JL, Pan PH, Thomas JA, Harris LC, D'Angelo R. A retrospective review of an epidural blood patch database: the incidence of epidural blood patch associated with obstetric neuraxial anesthetic techniques and the effect of blood volume on efficacy. Int J Obstet Anesth. 2017 Feb;29:10-17. doi: 10.1016/j.ijoa.2016.05.007. Epub 2016 Jun 3. PMID 27378709
- [Result] Safa-Tisseront V, Thormann F, Malassine P, Henry M, Riou B, Coriat P, Seebacher J. Effectiveness of epidural blood patch in the management of post-dural puncture headache. Anesthesiology. 2001 Aug;95(2):334-9. doi: 10.1097/00000542-200108000-00012. PMID 11506102
- [Result] Uppal V, Russell R, Sondekoppam R, Ansari J, Baber Z, Chen Y, DelPizzo K, Dirzu DS, Kalagara H, Kissoon NR, Kranz PG, Leffert L, Lim G, Lobo CA, Lucas DN, Moka E, Rodriguez SE, Sehmbi H, Vallejo MC, Volk T, Narouze S. Consensus Practice Guidelines on Postdural Puncture Headache From a Multisociety, International Working Group: A Summary Report. JAMA Netw Open. 2023 Aug 1;6(8):e2325387. doi: 10.1001/jamanetworkopen.2023.25387. PMID 37581893
- [Result] Mims SC, Tan HS, Sun K, Pham T, Rubright S, Kaplan SJ, Habib AS. Long-term morbidities following unintentional dural puncture in obstetric patients: A systematic review and meta-analysis. J Clin Anesth. 2022 Aug;79:110787. doi: 10.1016/j.jclinane.2022.110787. Epub 2022 Mar 28. PMID 35358942
- [Result] Ranganathan P, Golfeiz C, Phelps AL, Singh S, Shnol H, Paul N, Attaallah AF, Vallejo MC. Chronic headache and backache are long-term sequelae of unintentional dural puncture in the obstetric population. J Clin Anesth. 2015 May;27(3):201-6. doi: 10.1016/j.jclinane.2014.07.008. Epub 2014 Dec 4. PMID 25483233
- [Result] Heesen M, Klohr S, Rossaint R, Walters M, Straube S, van de Velde M. Insertion of an intrathecal catheter following accidental dural puncture: a meta-analysis. Int J Obstet Anesth. 2013 Jan;22(1):26-30. doi: 10.1016/j.ijoa.2012.10.004. Epub 2012 Dec 5. PMID 23219220
- [Result] Moschini V, Marra G, Dabrowska D. Complications of epidural and combined spinal-epidural analgesia in labour. Minerva Anestesiol. 2006 Jan-Feb;72(1-2):47-58. PMID 16407806
- [Result] Taivainen T, Pitkanen M, Tuominen M, Rosenberg PH. Efficacy of epidural blood patch for postdural puncture headache. Acta Anaesthesiol Scand. 1993 Oct;37(7):702-5. doi: 10.1111/j.1399-6576.1993.tb03793.x. PMID 8249562
- [Result] Headache Classification Committee of the International Headache Society (IHS) The International Classification of Headache Disorders, 3rd edition. Cephalalgia. 2018 Jan;38(1):1-211. doi: 10.1177/0333102417738202. No abstract available. PMID 29368949